CLINICAL TRIAL: NCT06047379
Title: An Open-label Phase 1/2 Dose Finding, Safety and Efficacy Study of Oral NEO212 in Patients With Astrocytoma IDH-mutant, Glioblastoma IDH-wildtype or Uncontrolled Brain Metastasis in Patients With Select Solid Tumors.
Brief Title: Safety and Efficacy of NEO212 in Patients With Astrocytoma IDH-mutant, Glioblastoma IDH-wildtype or Brain Metastasis
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Neonc Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEO212-01
Record Dates: First submitted 2023-08-17; First posted 2023-09-21 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Diffuse Astrocytoma, IDH-Mutant; Glioblastoma, IDH-wildtype; Brain Metastases, Adult; Cervical Cancer; Colorectal Cancer; Esophageal Cancer; Esophageal Squamous Cell Carcinoma; Gastric Cancer; Gastroesophageal Junction Adenocarcinoma; Head and Neck Squamous Cell Carcinoma; Melanoma; Merkel Cell Carcinoma; Microsatellite Instability-High Solid Malignant Tumor; Mismatch Repair Deficient Solid Malignant Tumor; Microsatellite Instability-High Colorectal Cancer; Mismatch Repair Deficient Colorectal Cancer; Non-small Cell Lung Cancer; Renal Cell Carcinoma; Small Cell Lung Cancer; Squamous Cell Carcinoma; Urothelial Carcinoma
Keywords: Astrocytoma; IDH-mutant; Glioblastoma; IDH-wildtype; Brain Metastases; CNS Tumor; GBM; NeOnc; Anova; NEO212; NEO100; TMZ
MeSH Terms: conditions — Astrocytoma; Glioblastoma; Brain Neoplasms; Uterine Cervical Neoplasms; Colorectal Neoplasms; Esophageal Neoplasms; Esophageal Squamous Cell Carcinoma; Stomach Neoplasms; Squamous Cell Carcinoma of Head and Neck; Melanoma; Carcinoma, Merkel Cell; Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Small Cell Lung Carcinoma; Carcinoma, Squamous Cell; Carcinoma, Transitional Cell; Central Nervous System Neoplasms | interventions — NEO212; Ipilimumab; pembrolizumab; Nivolumab; regorafenib; Carboplatin; Paclitaxel; IFL protocol; aflibercept; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Phase 2a Safety Run-In - NEO212 and Ipilimumab (Experimental): - Unresectable or metastatic melanoma with uncontrolled metastases to the brain.
  NEO212 - Starting one dose level under RP2D administered orally on days 1 - 5 of a 28-day treatment cycle, escalated to RP2D per Protocol dose escalation rules.
  Ipilimumab - 3 mg/kg administered IV over 90 minutes every 3 weeks for a maximum of 3 doses per package insert.
  Interventions: Drug: NEO212 Oral Capsule; Drug: Ipilimumab
- Phase 2a Safety Run-In - NEO212 and Pembrolizumab (Experimental): The following primary cancers with uncontrolled metrastases to the brain:
  * Unresectable or metastatic melanoma.
  * NSCLC expressing PD-L1, with no EGFR or ALK genomic tumor aberrations.
  * Metastatic NSCLC whose tumors express PD-L1.
  * EGFR or ALK genomic tumor aberrations must have disease progression.
  * SCLC.
  * Unresectable, recurrent HNSCC whose tumors express PD-L1.
  * HNSCC on or after platinum-containing chemotherapy.
  * Urothelial carcinoma whose tumors express PD-L1.
  * Urothelial carcinoma.
  * Microsatellite instability-high (MSI-H) or mismatch repair deficient (dMMR).
  * Microsatellite Instability-high or Mismatch Repair Deficient Colorectal Cancer (CRC).
  * Gastric or gastroesophageal junction adenocarcinoma.
  * Esophageal or gastroesophageal juncUon (GEJ).
  * Cervical cancer.
  * Merkel cell carcinoma.
  NEO212 - Same as Arm 1.
  Pembrolizumab - 200 mg administered every 3 weeks per package insert.
  Interventions: Drug: NEO212 Oral Capsule; Drug: Pembrolizumab
- Phase 2a Safety Run-In - NEO212 and Nivolumab (Experimental): The following primary cancers with uncontrolled metrastases to the brain:
  * Unresectable or metastatic melanoma.
  * Metastatic non-small cell lung cancer.
  * Advanced renal cell carcinoma.
  * Squamous cell carcinoma of the head and neck.
  * Urothelial carcinoma.
  * Microsatellite instability-high (MSI-H) or mismatch repair deficient (dMMR) colorectal cancer.
  * Unresectable esophageal squamous cell carcinoma (ESCC).
  NEO212 - Starting one dose level under RP2D administered orally on days 1 - 5 of a 28-day treatment cycle, escalated to RP2D per Protocol dose escalation rules.
  Nivolumab - 240 mg administered every 2 weeks per package insert
  Interventions: Drug: NEO212 Oral Capsule; Drug: Nivolumab
- Phase 2a Safety Run-In - NEO212 and Stivarga (Regorafenib) (Experimental): - Colorectal cancer (CRC) with uncontrolled metastases to the brain who have been previously treated with fluoropyrimidine-, oxaliplatin- and irinotecan-based chemotherapy, an anti-VEGF therapy, and, if KRAS wild type, an anU-EGFR therapy.
  NEO212 - Starting one dose level under RP2D administered orally on days 1 - 5 of a 28-day treatment cycle, escalated to RP2D per Protocol dose escalation rules.
  Stivarga - 160 mg orally, once daily for the first 21 days of each 28-day cycle per package insert
  Interventions: Drug: NEO212 Oral Capsule; Drug: Regorafenib
- Phase 2a Safety Run-In - NEO212 and CarbolaUn (ParaplaUn) + Paclitaxel (Taxol) (Experimental): - Colorectal cancer (CRC) with uncontrolled metastases to the brain.
  NEO212 - Starting one dose level under RP2D administered orally on days 1 - 5 of a 28-day treatment cycle, escalated to RP2D per Protocol dose escalation rules.
  Carboplatin - 300 mg/m2 IV on day 1 every 4 weeks for 6 cycles per package insert.
  Paclitaxel - 135mg/m2 IV administered over 24 hours, every 3 weeks per package insert.
  Interventions: Drug: NEO212 Oral Capsule; Drug: Carboplatin; Drug: Paclitaxel
- Phase 2a Safety Run-In - NEO212 and FOLFIRI (Zaltrap) + Bevacizumab (Avastin) (Experimental): - Metastatic colorectal cancer (mCRC) with uncontrolled metastases to the brain, that is resistant to or has progressed following an oxaliplatin-containing regimen
  NEO212 - Starting one dose level under RP2D administered orally on days 1 - 5 of a 28-day treatment cycle, escalated to RP2D per Protocol dose escalation rules.
  FOLFIRI - 4 mg/kg aIV over 1 hour every 2 weeks.
  Bevacizumab - 10 mg/kg IV every 2 weeks.
  Interventions: Drug: NEO212 Oral Capsule; Drug: FOLFIRI Protocol; Drug: Bevacizumab
- Phase 2b efficacy - NEO212 for Astrocytoma IDH-mutant and Glioblastoma IDH-wildtype (Experimental): Patients receiving NEO212 alone for treatment of Astrocytoma IDH-mutant and Glioblastoma IDH-wildtype.
  NEO212 - Starting one dose level under RP2D administered orally on days 1 - 5 of a 28-day treatment cycle, escalated to RP2D per Protocol dose escalation rules.
  Interventions: Drug: NEO212 Oral Capsule
- Phase 2b efficacy - NEO212 & SOC for Uncontrolled Metastases to the Brain (Experimental): Patients receiving NEO212 in combination with select standard of care treatments for treatment of uncontrolled metastases to the brain.
  NEO212 - Starting one dose level under RP2D administered orally on days 1 - 5 of a 28-day treatment cycle, escalated to RP2D per Protocol dose escalation rules.
  SOC treatments established to be safe in Phase 2a of the study will be used in this arm of Phase 2b.
  Interventions: Drug: NEO212 Oral Capsule; Drug: Ipilimumab; Drug: Pembrolizumab; Drug: Nivolumab; Drug: Regorafenib; Drug: Carboplatin; Drug: Paclitaxel; Drug: FOLFIRI Protocol; Drug: Bevacizumab

INTERVENTIONS:
Drug: NEO212 Oral Capsule — NEO212 is a novel chemical entity that was generated by covalent conjugation of temozolomide (TMZ) with perillyl alcohol (POH).
  Other Names: POH-TMZ
Drug: Ipilimumab — Ipilimumab, sold under the brand name Yervoy, is a monoclonal antibody medication that works to activate the immune system by targeting CTLA-4, a protein receptor that downregulates the immune system. Cytotoxic T lymphocytes can recognize and destroy cancer cells.
  Other Names: Yervoy
  Arms: Phase 2a Safety Run-In - NEO212 and Ipilimumab; Phase 2b efficacy - NEO212 & SOC for Uncontrolled Metastases to the Brain
Drug: Pembrolizumab — Pembrolizumab, sold under the brand name Keytruda, is a humanized antibody used in cancer immunotherapy that treats melanoma, lung cancer, head and neck cancer, Hodgkin lymphoma, stomach cancer, cervical cancer, and certain types of breast cancer. It is given by slow injection into a vein.
  Other Names: Keytruda
  Arms: Phase 2a Safety Run-In - NEO212 and Pembrolizumab; Phase 2b efficacy - NEO212 & SOC for Uncontrolled Metastases to the Brain
Drug: Nivolumab — Nivolumab, sold under the brand name Opdivo, is a medication used to treat a number of types of cancer.
  Other Names: Opdivo
  Arms: Phase 2a Safety Run-In - NEO212 and Nivolumab; Phase 2b efficacy - NEO212 & SOC for Uncontrolled Metastases to the Brain
Drug: Regorafenib — Regorafenib, sold under the brand name Stivarga among others, is an oral multi-kinase inhibitor developed by Bayer which targets angiogenic, stromal and oncogenic receptor tyrosine kinase. Regorafenib shows anti-angiogenic activity due to its dual targeted VEGFR2-TIE2 tyrosine kinase inhibition
  Other Names: Stivagra
  Arms: Phase 2a Safety Run-In - NEO212 and Stivarga (Regorafenib); Phase 2b efficacy - NEO212 & SOC for Uncontrolled Metastases to the Brain
Drug: Carboplatin — Carboplatin, sold under the trade name Paraplatin among others, is a chemotherapy medication used to treat a number of forms of cancer. This includes ovarian cancer, lung cancer, head and neck cancer, brain cancer, and neuroblastoma. It is used by injection into a vein.
  Other Names: Paraplatin
  Arms: Phase 2a Safety Run-In - NEO212 and CarbolaUn (ParaplaUn) + Paclitaxel (Taxol); Phase 2b efficacy - NEO212 & SOC for Uncontrolled Metastases to the Brain
Drug: Paclitaxel — Paclitaxel, sold under the brand name Taxol among others, is a chemotherapy medication used to treat ovarian cancer, esophageal cancer, breast cancer, lung cancer, Kaposi's sarcoma, cervical cancer, and pancreatic cancer. It is administered by intravenous injection
  Other Names: Taxol
  Arms: Phase 2a Safety Run-In - NEO212 and CarbolaUn (ParaplaUn) + Paclitaxel (Taxol); Phase 2b efficacy - NEO212 & SOC for Uncontrolled Metastases to the Brain
Drug: FOLFIRI Protocol — FOLFIRI is a chemotherapy regimen for treatment of colorectal cancer. It is made up of the following drugs:
  FOL - folinic acid (leucovorin), a vitamin B derivative with multiple applications, which in this context increases the cytotoxicity of 5-fluorouracil; F - fluorouracil (5-FU), a pyrimidine analog and antimetabolite which incorporates into the DNA molecule and stops synthesis; and IRI - irinotecan (Camptosar), a topoisomerase inhibitor, which prevents DNA from uncoiling and duplicating.
  Other Names: Zaltrap
  Arms: Phase 2a Safety Run-In - NEO212 and FOLFIRI (Zaltrap) + Bevacizumab (Avastin); Phase 2b efficacy - NEO212 & SOC for Uncontrolled Metastases to the Brain
Drug: Bevacizumab — Bevacizumab, sold under the brand name Avastin among others, is a medication used to treat a number of types of cancers and a specific eye disease. For cancer, it is given by slow injection into a vein and used for colon cancer, lung cancer, glioblastoma, and renal-cell carcinoma
  Other Names: Avastin; Mvasi; Zirabev; Alymsys; Vegzelma
  Arms: Phase 2a Safety Run-In - NEO212 and FOLFIRI (Zaltrap) + Bevacizumab (Avastin); Phase 2b efficacy - NEO212 & SOC for Uncontrolled Metastases to the Brain

SUMMARY:
This multi-site, Phase 1/2 clinical trial is an open-label study to identify the safety, pharmacokinetics, and efficacy of a repeated dose regimen of NEO212 alone for the treatment of patients with radiographically-confirmed progression of Astrocytoma IDH- mutant, Glioblastoma IDH-wildtype, and the safety, pharmacokinetics and efficacy of a repeated dose regimen of NEO212 when given with select SOC for the treatment of solid tumor patients with radiographically confirmed uncontrolled metastases to the brain.

The study will have three phases, Phase 1, Phase 2a and Phase 2b.

DETAILED DESCRIPTION:
This multi-site, Phase 1/2 clinical trial is an open-label study to identify the safety, pharmacokinetics, and efficacy of a repeated dose regimen of NEO212 for the treatment of patients with radiographically-confirmed progression of Astrocytoma IDH-mutant, Glioblastoma IDH-wildtype, and the safety, pharmacokinetics and efficacy of a repeated dose regimen of NEO212 when given with select SOC for the treatment of solid tumor patients with radiographically confirmed uncontrolled brain metastasis. The study will have three phases, Phase 1, Phase 2a and Phase 2b.

Phase 1 is a standard cohort dose escalation 3+3 design with a modified Fibonacci dose escalation used to determine the maximum tolerated dose to select a recommended Phase 2 dose (RP2D) of NEO212 for Phase 2a and Phase 2b. The initial dose of NEO212 will be 170 mg and the dose will increase in successive cohorts (220, 400, 610, 810, and 1,000 mg) until a MTD is reached and a RP2D is selected. There will be up to 42 patients enrolled in Phase 1. In the event two DLTs are experienced in any cohort, a dose de- escalation cohort will be followed (with half of the dose increase from the previous cohort) to determine the MTD/RP2D.

Phase 2a is a safety run-in study with a standard 3+3 design used to confirm the safety of the MTD/RP2D of NEO212 when given in combination with select SOC regimens for patients with uncontrolled metastases to the brain. There will be up to 12 patients enrolled into each combination regimen to confirm safety. One dose below the NEO212 MTD/RP2D Cohort Dose will be administered as a starting dose to establish safety (3+3), before moving to Phase 2b with the MTD/RP2D (3+3). In the event that two DLTs are experienced for patients receiving the MTD/RP2D in combination with SOC, the dose de-escalation cohort will be expanded to determine the MTD for a newly established Phase 2b Treatment Group.

Phase 2b is a dose expansion study to assess efficacy of NEO212 alone, at the MTD/RP2D in patients with Astrocytoma IDH-mutant, Glioblastoma IDH-wildtype as a single Treatment Group. A second Treatment Group to study the MTD/RP2D of NEO212 in combination with select SOC regimens in patients with solid tumors and uncontrolled metastases to the brain established in Phase 2a will be evaluated. Phase 2b will be initiated for patients with Astrocytoma IDH-mutant or Glioblastoma IDH-wildtype alongside Phase 2a. There will be up to 28 patients enrolled to have 27 evaluable patients enrolled in each Phase 2b Treatment Group.

For all phases of the study, NEO212 will be self-administered daily for days 1-5 of a 28- day treatment cycle.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be ≥ 18yrs of age.
* Patient must have the ability to understand, and the willingness to sign, a written informed consent form.
* Patient has been on a stable or decreasing dose of steroids for at least five days prior to the date of informed consent.
* Any toxicity from prior therapy must be resolved or at maximum Grade 1 prior to initiation of NEO212.
* If progression of disease occurs within 90 days or conformal radiation, the progression/recurrence must be outside of the radiation field or proven by biopsy/resection.
* Patient with Astrocytoma IDH-mutant, Glioblastoma IDH-wildtype must have a Karnofsky Performance Status (KPS) of ≥ 60.
* Patient with select solid tumors must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Patient must have an expected survival or at least three months.
* Patient must have a baseline MRI of the brain with gadolinium within 14 days of administration of NEO212.
* Patient with select solid tumors must have a baseline CT scan with IV contrast and oral contrast of neck, chest, abdomen and pelvis within 14 days of administration of NEO212.
* Patients must be able to comply with all study assessments.
* If patient suffers from seizures (s)he must be controlled on a stable dose of anti-epileptics for 14-days prior to the date of informed consent.
* Patient must have adequate organ and marrow function as follows:

  * Absolute neutrophil count ≥ 1,500/microliter
  * Platelets ≥ 100,000/microliter
  * Total bilirubin within normal institutional limits
  * AST (SGOT) / ALT (SPGT) ≤ 2.5 x institutional upper limit of normal
  * Creatinine clearance (CrCl) of >60 mL/min (using the Cockcroft-Gault formula or 24- hour urine collection).
* Female patients of child-bearing potential and male patients must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for 30 days prior to the first dose of NEO212, for the duration of study participation, and for 90 days following completion of therapy.

A female of child-bearing potential is any women (regardless of sexual orientation, not having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

* Has not undergone a hysterectomy or bilateral oophorectomy; or
* Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has not had menses at any time in the preceding 12 consecutive months).
* A negative serum pregnancy test will be required of all female patients of child-bearing potential within seven days prior to the receipt of NEO212.
* A serum pregnancy test will be repeated immediately if pregnancy is suspected.

Phase 1: (dose escalation)

* Patient must:

  * have radiographically confirmed Astrocytoma IDH-mutant, Glioblastoma IDH-wildtype following previous radiation therapy or treatment with temozolomide and radiation, or
  * have select solid tumors with uncontrolled metastases to the brain (confirmed by cranial CT or MRI) that is not controlled by surgery or radiation therapy and receiving one of the protocol approved SOC regimens.
* Patients receiving prior systemic therapy must have a minimum wash-out period (defined as the period prior to receipt of the first dose of NEO212) of:

  * 28 days or 5 half-lives (whichever is shorter) elapsed from the administration from any experimental agent;
  * 2 weeks from administration of immunotherapies;
  * 28 days from administration of cytotoxic agents; and
  * 7 days from administration of non-cytotoxic agents (interferon, tamoxifen, thalidomide, cis-retinoic acid, and herbal medicine).

NOTE: No washout is necessary for alternating electrical fields.

Phase 2a: (safety run-in)

* Patient must have select solid tumors with uncontrolled metastases to the brain (confirmed by cranial CT or MRI) that is not controlled by surgery or radiation therapy and receiving one of the protocol approved SOC regimens.
* Patients receiving prior systemic therapy must be receiving one of the protocol approved Standard of Care (SOC) regimens.
* Patient must have measurable/evaluable CNS disease per RANO or RANO-BM criteria.
* Patient must have measurable/evaluable systemic disease per RECIST v1.1 criteria.

Phase 2b: (efficacy)

* Patient must:

  * have radiographically confirmed Astrocytoma IDH-mutant, Glioblastoma IDH-wildtype following previous radiation therapy or treatment with temozolomide and radiation, or
  * have select solid tumors with uncontrolled metastases to the brain (confirmed by cranial CT or MRI) that is not controlled by surgery or radiation therapy and receiving one of the protocol approved SOC regimens.
* Patients receiving prior systemic therapy must be receiving one of the protocol approved Standard of Care (SOC) regimens.
* Patient must have measurable/evaluable CNS disease per RANO or RANO-BM criteria
* Patient with select solid tumors must have measurable/evaluable systemic disease per RECIST v1.1 criteria.
* Creatinine clearance (CrCl) of >60 mL/min (using the Cockcroft-Gault formula or 24-hour urine collection). Female patients of child-bearing potential and male patients must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for 30 days prior to the first dose of NEO212, for the duration of study participation, and for 90 days following completion of therapy.

Exclusion Criteria: (all Phases)

* Patient in Phase 1 concurrently receiving any other antitumor therapy.
* Patient in Phase 2a or 2b who is concurrently receiving any SOC therapy not listed in Appendix 1.
* Patients with metastases to the spinal cord parenchyma.
* Patients with metastases to the meninges.
* Patient has received stereotactic or highly conformal radiotherapy to CNS lesions within 2 weeks before receipt of NEO212.
* Patient with history of known leptomeningeal involvement.
* Patient has prior history or new diagnosis of secondary cancer within five years prior to the date of informed consent, except for basal cell carcinoma or squamous cell carcinoma of the skin.
* Patient has a corrected QT interval (using Fridericia's correction formula) (QTcF) of >470 msec, a history of additional risk factors for TdP (e.g. heart failure, hypokalemia), and/or the use of concomitant medications that prolong QT/QTc interval.
* Patient had surgery within 7 days prior to the date of informed consent.
* Patient has not recovered to Grade 1 from treatment related adverse events due to chemotherapy, immunotherapy, or radiation therapy.
* Patient had prior treatment with perillyl alcohol.
* Patient has a history of allergic reactions attributed to perillyl alcohol.
* Patients in Phase 2b with Astrocytoma IDH-mutant, or Glioblastoma IDH-wildtype who have had more than one recurrence or progression of his/her primary CNS tumor(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1: safety and tolerability of increasing dose levels of orally administered NEO212 alone in patients with Astrocytoma IDH-mutant, Glioblastoma IDH-wildtype or patients with select solid tumors with uncontrolled metastases to the brain | 6 months
  As determined by incidence and severity of adverse events according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v5.0
Phase 1: Identify the maximum tolerated dose (MTD) of NEO212 | 6 months
  Maximum Tolerated Dose of NEO212 as determined by the dose escalation rules.
Phase 1: Determine the recommended Phase 2 dose (RP2D) of NEO212 | 6 months
  Determine the recommended Phase 2 dose (RP2D) of NEO212
Phase 2a: Assess the safety and tolerability of orally administered NEO212 in combination with select SOC regimens following a standard 3+3 design in patients with select solid tumors with uncontrolled metastases to the brain | 6 months
  Determined by incidence and severity of adverse events determined according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE v5.0).
Phase 2b: Determine the intracranial progression-free survival rate at six months (PFS6) of orally administered NEO212 alone in patients with Astrocytoma IDH-mutant, Glioblastoma IDH-wildtype. | 6 months
  Determine the intracranial progression-free survival rate at six months (PFS6) of orally administered NEO212 alone in patients with Astrocytoma IDH-mutant, Glioblastoma IDH-wildtype.
Phase 2b: Determine the intracranial progression-free survival rate at six months (PFS6) of orally administered NEO212 in combination with select SOC regimens in patients with select solid tumors with uncontrolled metastases to the brain. | 6 months
  Determine the intracranial progression-free survival rate at six months (PFS6) of orally administered NEO212 in combination with select SOC regimens in patients with select solid tumors (see Appendix 2) with uncontrolled metastases to the brain.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Chen, MD, PhD, Study Chair — NeOnc Technologies; Josh Neman, PhD, Study Director — NeOnc Technologies Holdings, Inc.
Locations (5):
- United States (5):
  - Precision NextGen Oncology, Beverly Hills, California
  - OPN Healthcare, Inc, Glendale, California
  - University of Southern California, Los Angeles, California
  - Baylor, Scott and White Research Institute, Dallas, Texas
  - Northwest Medical Specialties, Tacoma, Washington